CLINICAL TRIAL: NCT01204424
Title: Klinische Prüfung Zur Untersuchung Der Sicherheit Und Machbarkeit Des Crestalen, Minimal-invasiven Kieferknochenaufbaus (Sinuslift) Mit Der Druck-kammerknochenfräse (DDK) Und Der Sinusvibrationspumpe (SVP)
Brief Title: Clinical Investigation to Assess the Safety and Feasibility of the Crestal, Minimal-invasive Sinus Floor Augmentation With the Pressure Chamber Drill (DKK) and the Sinus Vibration Pump (SVP)
Acronym: DKK SVP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeder GmbH (Industry)
Responsible Party: Andreas Bayerle, CEO, JEDER GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKK-SVP-10 Prot. 1.4; EK_10_101_0610 (Other: Ethikkommission-Vienna-Austria-Europe:)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Insufficient Bone Mass in the Maxilla for Dental Implants
Keywords: minimal invasive; sinus floor augmentation; sinuslift; dental implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: minimal-invasive sinus floor augmentation with the DKK and SVP (JEDER Syst.) — minimal-invasive sinus floor augmentation with the DKK and SVP (JEDER Syst.)
Device: minimal invasive crestal sinus lift with the JEDER Systh. — The mucous membrane is opened from the toothless part of the maxillary crest up to the bone and the bone is scraped by a cylindrical cutter in the shape of a tunnel up to slightly underneath the maxillary sinus membrane and hydraulic pressure is being built up within the DKK. A centrally placed drill within the DKK slowly moves in the direction of the membrane. At the moment of the first minimal perforation of the remaining bone the pressurized fluid pushes the membrane back and ensures that the membrane is not perforated by the drill.
  The SVP is used to generate hydraulic vibrations, which help to further raise the membrane from the bone (principle of the "percussion drill"). After the maxillary sinus membrane has successfully been elevated, the working fluid is extracted and bone replacement material is introduced via the bore.
  Other Names: minimal invasive crestal sinuslift

SUMMARY:
The success of dental implants is based on a variety of factors including; surgical technique, health of the patient, operator skill and, to a significant part, sufficient bone for the placement and integration of dental implants. To that end, the replacement of the maxillary posterior teeth have presented a considerable challenge because, after the loss of maxillary posterior teeth the quality and quantity of the remaining supporting bone may be insufficient to support implants properly or reliably. To overcome the deficiency of insufficient vertical bone mass of the maxilla, several surgical techniques have been developed to increase available bone mass for the replacement of dental implants by bone augmentation.

The conventional procedure for a sinus lift (Caldwell-Luc procedure) requires preparation of a mucoperiosteal flap in the buccal molar region and to cut an oval window in the thus exposed bone, without damage to the subjacent maxillary sinus membrane. The procedure is very invasive and subjects the patient to great stress as a result of substantial swelling and discoloration of up to 10 days, and possibly of pain. This surgical procedure is oftentimes referred to as "open" or "classic" sinus lift. This technique is fraught with many risks and complications because of the limitations of healing potential in the maxillary sinus. In spite of these risks many patients undergo this procedure because of the strong desire to replace missing maxillary teeth with dental implants.

An alternative approach to the maxillary sinus from the inferior approach of the alveolar ridge utilizing solid cylindrical osteotomes was described by Dr. Summers (crestal sinus lift). It is a more conservative approach and is less invasive. It was developed to eliminate the risks described above.While this technique is safer, an overzealous use of an osteotome during the placement of the regenerative material can result in the perforation of the subantral membrane with disadvantages discussed above.

Dr. Eder has developed an innovative way - the JEDER System - of carrying out a crestal sinus lift that substantially reduces the risk of perforating the subantral membrane. This minimal- invasive way uses 2 newly developed and successfully patented instruments, the "Druckkammerknochenfräse" DKK and the "Sinusvibrationspumpe" SVP. Following JEDER Syst. the mucous membrane of the mouth is opened from the toothless part of the maxillary crest up to the bone and the bone is scraped by a cylindrical cutter in the shape of a tunnel up to slightly underneath the maxillary sinus membrane.

The aim of the study is to assess the efficacy and safety of the JEDER Syst., which was already demonstrated in 50 treatment attempts. The results of this study will be used for the certification process to enable the declaration of conformity for the market approval.

The main outcome parameter is the perforation rate of the subantral membrane intraoperatively and within 6 weeks after the operation.

Risk benefit assessment:

In the present study there will be no additional examinations undertaken compared to patients which undergo the conventional procedure. The conventional procedure is associated with a risk of membrane perforation and consecutive diseases like infection, swelling and pain. All these inconveniences should be avoided by using the JEDER Syst. If the worst case scenario - the perforation of the subantral membrane - happens, the conventional method will be used. Therefore, the risk-benefit assessment

ELIGIBILITY:
Inclusion Criteria:

* demand for sinus floor elevation (regio 4 to 7)
* loss of teeth (regio 4 to 7)
* needed extraction of teeth (regio 4 to 7)

Exclusion Criteria:

* maxillary bone mass <3mm
* severe chronic illness or immune deficiency
* cortisone therapy
* sinus membrane membrane hight >5mm
* chronic sinusitis
* smoking >20 Zigarettes
* missing dental hygiene

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
perforation rate of the subantral membrane in the sinus maxillaris | intraoperativ and within 6 weeks after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Michaela M Bayerle-Eder, Prof., MD, MBA, Study Director — Medical University Vienna, Vienna Austria, Europe
Locations (1):
- Ordination Dr. Klaus Eder, Vienna, Vienna, Austria